CLINICAL TRIAL: NCT05613114
Title: Effect of Dalfampridine in Patients With Hereditary Spastic Paraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Ferda Selcuk, Assist Prof. Dr., European University of Lefke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 45/20
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — 4-Aminopyridine; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication (Experimental): Dalfampridine plus physiotherapy
  Interventions: Drug: Dalfampridine 10 MG; Behavioral: Physiotherapy
- No Medication (Placebo Comparator): Placebo plus physiotherapy
  Interventions: Drug: Placebo; Behavioral: Physiotherapy

INTERVENTIONS:
Drug: Dalfampridine 10 MG — The participants in the experimental group received dalfampridine administered as 10 mg extended-release tablets every twelve hours for 8 weeks.
  Arms: Medication
Drug: Placebo — Control group received a placebo drug with the same administration method (2 times per week for the total duration of 8 weeks).
  Arms: No Medication
Behavioral: Physiotherapy — Conventional physiotherapy program including stretching and flexibility, strengthening, walking and balance exercises which were mainly focused on the lower limbs and improving walking. The program was applied 2 times per week for the total duration of 8 weeks.

SUMMARY:
There are limited but encouraging results supporting the use of dalfampridine in patients with hereditary spastic paraplegia. The investigators aimed to investigate the effects of dalfampridine on walking speed, muscle length, spasticity, functional strength, and functional mobility in patients with hereditary spastic paraplegia. In this triple-blinded, randomized, placebo-controlled trial, 4 patients with hereditary spastic paraplegia received dalfampridine (10 mg twice daily) plus physiotherapy (2 times per week), and 4 patients received placebo plus physiotherapy for a total duration of 8 weeks. The assessor and treating physiotherapists, and patients were masked to the group allocation. The primary outcome was Timed 25-foot Walk Test at the end of the 8-week treatment. The secondary outcome measures were functional mobility, functional muscle strength, muscle length, and spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hereditary Spastic Paraplegia at least 1 year ago

Exclusion Criteria:

* Having another neurological disorder
* An orthopedic deformity in the lower extremity
* Having a serious cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Timed 25-foot Walk Test | Change from baseline to week 8
  The Timed 25-foot walk test (T25FW) is considered the "best characterized objective measure of walking disability and can be used across a wide range of walking disabilities". For the T25-FW, patients were instructed to walk as fast as they could in a safemanner along amarked 25-foot course. The time in seconds to complete each test was recorded, and the test was immediately repeated.

SECONDARY OUTCOMES:
Sit to Stand Test | Change from baseline to week 8
  30 second Chair-Stand Test which is a reliable and valid measure used to assess lower extremity strength and endurance is used where the number of sitting and getting up within 30 seconds gives the score of the test.
Timed Up and Go test | Change from baseline to week 8
  Functional mobility was evaluated using the Timed up and Go Test 'TUG' test, which is also reliable and valid test for people with Parkinson's disease. (Morris2001; Van2016). Upon issuing the command "Go," the participants stood up from a normal chair, walked 3 meters, turned, walked back to the chair, and sat. The time began with the command "Go" and ended when the participants sat back to the chair. This test was repeated three times, and the shortest performance time was recorded
Modified Ashworth Scale | Change from baseline to week 8
  Modified Ashworth Scale (MAS) is one of the reliable and valid methods to measure muscle spasticity. The procedure to evaluate specific muscle groups; passively moved through the range of motion of a limb, and the resistance encountered during muscle stretch is rated on a five-point scale. Ashworth defines this rating as; 0 = no increase in tone, 1 = slight increase in tone at the end of the range of motion, 1+ = slight increase in tone throughout less than half the range of motion, 2 = increased muscle tone throughout the full range of motion, but passive movement is present. 3=tone movement that makes passive movement difficult, 4=rigidity .
Muscle Length Measurement | Change from baseline to week 8
  Bilateral muscle length measurements were obtained using a standard goniometer. The patient positioned in supine position; the dorsiflexion has been tested for the gastrocnemius, the straight leg rise - hip angle has been measured to assess hamstrings, the Thomas test was used to assess iliopsoas and hip abduction angle was used for adductor group muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Ferda Selcuk, Principal Investigator — European University of Lefke
Locations (1):
- Dr. Burhan Nalbantoğlu State Hospital, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selcuk Muhtaroglu F, Belgen Kaygisiz B, Usar Incirli S, Kahraman T. Dalfampridine as a promising agent in the management of hereditary spastic paraplegia: A triple-blinded, randomized, placebo-controlled pilot trial. J Clin Neurosci. 2023 Nov;117:136-142. doi: 10.1016/j.jocn.2023.09.026. Epub 2023 Oct 5. PMID 37804674